CLINICAL TRIAL: NCT06531889
Title: Core Stabilization Exercises in Shoulder Impingement Syndrome: A Preliminary Retrospective Study
Brief Title: Core Stabilization Exercises on Shoulder Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Collaborators: Yeditepe University (Other)
Responsible Party: Principal Investigator, Nuray Alaca, Assoc. Prof Nuray Alaca, Acibadem University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 37068608-6100-15-1757
Record Dates: First submitted 2023-12-15; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Subacromial Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- classical physiotherapy program (Active Comparator): The group in classical physiotherapy program; n=25 (3 days per week for six weeks)
  Interventions: Other: classical physiotherapy program
- core stabilization group (Experimental): The group in which core stabilization was also performed in addition to classical physiotherapy program; n=25 (3 days per week for 6 weeks)
  Interventions: Other: classical physiotherapy program; Other: Core Stabilization Exercises

INTERVENTIONS:
Other: classical physiotherapy program — Classical physiotherapy program=Classical physiotherapy program included transcutaneous electrical nerve stimulation, infrared radiation for 15 min, continuous ultrasound for 5 min and home exercise program. For active assistive shoulder range of motion (ROM), home exercises included the Codman exercise, flexion exercise at the ladder, and the Wand exercise, as well as some strengthening and stretching exercises performed at the pain limit with 10 repetitions twice a day (six weeks)
Other: Core Stabilization Exercises — The interventions of the core exercise were applied when the patient lay on his/her back with his/her knees at flexion. The number of repeats for each exercise was five, and these exercises were done 3 times a week for 6 weeks with the same physiotherapist. The further steps in the exercises were extended according to the activation duration of the core muscles, and this extension was elongated 5 s
  Arms: core stabilization group

SUMMARY:
The objective of this retrospective study was to look into the effects of core stabilization exercises applied in conjunction with classic physiotherapy program on pain, muscle strength, disability, and posture in SIS.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 35 and 60 who were diagnosed by a Physical Therapy and Rehabilitation doctor with at least ten years of experience, whose SIS was confirmed by MRI, and who had shoulder complaints for at least three months, patients with positive signs, a positive Hawkins-Kennedy test, significant loss of active and passive shoulder movements or painful range of motion (ROM), and patients whose treatment and evaluation methods were appropriate for the study design were enrolled in the study

Exclusion Criteria:

* Patients who had upper extremity surgery, patients with a history of shoulder trauma and corticosteroid application to the shoulder region in the previous year, a history of shoulder dislocation, infection, tumor, adhesive capsulitis, reflex sympathetic dystrophy, congenital anomaly, rheumatic disease, and chronic severe systemic disease, as well as professional athletes and patients whose evaluations were missing in the previous month were excluded

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
The Numerical Rating Scale (NPRS-11) | Change from baseline pain score at 6th week
  The Numerical Rating Scale (NPRS-11) is an 11-point scale for self-report of pain. It is the most commonly used unidimensional pain scale. The respondent selects a whole number (integers 0-10) that best reflects the intensity (or other quality if requested of his/her pain.0 point is the minimum and 10 point is the maximum. The higher the score, the more severe the pain.
New York Posture Rating Method to determine their postures | Change from baseline pain score at 6th week
  The rating chart is used to assess 13 areas of the body, based on the assumption that posture is the alignment of the body and its segments. 13 regions (head, neck, shoulder, scapula, upper thoracic, waist, rips, abdomen, hips, knees, legs, feet and toes) are assessed in two different positions (lateral and posterior). A score is allocated to each area according to the position: 5 points to the correct position; 3 points for a slight deviation, and 1 point for a pronounced deviation. Total score is between 18-90 points. higher the points better the postural alignment
Shoulder pain and disability index | Change from baseline score of The Shoulder Pain and Disability Index at 6th week
  The Shoulder Pain and Disability Index (SPADI) was developed to measure current shoulder pain and disability in an outpatient setting. The SPADI contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability between 0 to 100, with a higher value indicating worse condition.

SECONDARY OUTCOMES:
Shoulder mobility on the Shoulder Range of Motion | Change from baseline range of motion at 6th week
  Shoulder ROM was measured in six directions (Flexion, Extension, Abduction, Adduction, Right rotation, Left rotation) with goniometer.
Core muscle strength test | Change from baseline strenght score at 6th week
  The level of difficulty was raised from stage 1 to stage 5. high values are indicative of positive progress
Endurance of Core Muscles | Change from baseline endurance score at 6th week
  Each test was repeated three times, and the average of the measurements was used. The Biering-Sørensen test measures how many seconds the participant can keep the unsupported upper part of the body in a horizontal position.high values are indicative of positive progress
Manual muscle test | Change from baseline manual muscle testing score at 6th week
  The lowest value is zero and the highest value is 5. high values are indicative of positive progress

CONTACTS AND LOCATIONS:
Overall Officials: Nuray ALACA, Study Director — Acibadem University
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided